CLINICAL TRIAL: NCT02742168
Title: Clinical Study of 99mTc-3PRGD2 SPECT/CT in Diagnosis and Efficacy Evaluation of Breast Cancer
Brief Title: 99mTc-3PRGD2 SPECT/CT in Breast Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Fujian Medical University (Other)
Responsible Party: Principal Investigator, Weibing Miao, PhD, Director, Department of Nuclear Medicine, First Affiliated Hospital of Fujian Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FirstAHFujian2
Record Dates: First submitted 2016-03-08; First posted 2016-04-18 (Estimated); Last update posted 2020-08-03 (Actual); Status verified 2020-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: The participants were underwent the 99mTc-3PRGD2 imaging and 18F-FDG imaging within one week.
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Breast Cancer,99mTc-3PRGD2,SPECT/CT (Experimental): Determine if 99mTc-3PRGD2 SPECT/CT is safe and effective in diagnosis and efficacy evaluation of breast cancer
  Interventions: Radiation: 99mTc-3PRGD2

INTERVENTIONS:
Radiation: 99mTc-3PRGD2 — Diagnostic group：For patients in suspicion of breast cancer, single intravenous bolus injection of nearly 0.3 mCi/kg body weight of 99mTc-3PRGD2 on day one of the treatment period, whole-body planar and lesions SPECT/CT to determine the accumulation of 99mTc-3PRGD2 in the tumors and the other parts of the body.
  Efficacy evaluation group：patients firstly diagnose with malignant lesions ,and prepare to chemotherapy(including neoadjuvant chemotherapy) or radiotherapy.the same dose of 99mTc-3PRGD2 will be intravenously injected into the patients before treatment ,the second period,the sixth period( almost three months after the initial treatment)，whole-body planar and lesions SPECT/CT to assess the value of 99mTc-3PRGD2 in evaluation of cancers.
  Other Names: 99mTc-HYNIC-3PRGD2

SUMMARY:
This is an open-label SPECT/CT (single photon emission computed tomography / computed tomography) study to investigate clinical study of 99mTc-3PRGD2 SPECT/CT in diagnosis and efficacy evaluation of breast cancer. Diagnostic group: for patients in suspicion of breast cancer. The standard of truth for diagnosis was based on histopathologic findings after surgical removal of the tumor or a definite diagnosis from fine needle aspiration biopsy. A single dose of nearly 0.3 mCi/kg (milli-Curie/kilogram) body weight of 99mTc-3PRGD2 ( ≤ 20 µg 3PRGD2) will be intravenously injected into the patients. Visual and semiquantitative method will be used to assess the whole-body planar and lesions SPECT/CT images.

Efficacy evaluation group: for patients firstly diagnose with malignant tumors (breast cancer), and prepare to chemotherapy(including neoadjuvant chemotherapy) or radiotherapy. The standard of truth for diagnosis was based on histopathologic findings after fine needle aspiration biopsy. A single dose of nearly 0.3 mCi/kg body weight of 99mTc-3PRGD2 ( ≤ 20 µg 3PRGD2) will be intravenously injected into the patients before treatment, the second period, sixth period. Visual,semiquantitative method will be used to assess the whole-body planar and lesions SPECT/CT images. By comparing with result of the other related imaging, for instance, PET/CT (positron emission tomography/computed tomography), CT (computed tomography), MRI (magnetic resonance imaging), Doppler Ultrasound, Mammography, etc.

DETAILED DESCRIPTION:
Integrin αvβ3 is an important member of integrin receptor family and expressed preferentially on the activated endothelial cells of angiogenesis and some types of tumor cells, but not or very low on the quiescent vessel cells and other normal cells. Therefore, the integrin αvβ3 receptor is becoming a valuable target for diagnosis and response evaluation of malignant tumors.

The tri-peptide sequence of arginine-glycine-aspartic acid (RGD) can specifically bind to the integrin αvβ3 receptor. Accordingly, a variety of radiolabeled RGD-based peptides have been developed for non-invasive imaging of integrin αvβ3 expression via single photon emission computed tomography (SPECT)or positron emission tomography (PET). Among all the RGD radiotracers studied, several RGD monomers have been investigated in clinical trials, and the preliminary results demonstrated specific imaging of various types of tumors, and the tumor uptake correlated well with the level of integrin αvβ3 expression. Recently, several RGD dimeric peptides with PEG linkers have been studied. The new types of RGD peptides showed much higher in vitro integrin αvβ3-binding affinity than the single RGD tri-peptide sequence, and importantly, they exhibited significantly increased tumor uptake and improved in vivo kinetics in animal models. As a representative, 99mTc-3PRGD2 could be easily prepared and exhibited excellent in vivo behaviors in animal models. No adverse reactions are observed in animal models to date.

For the further interests in clinical trial of 99mTc-3PRGD2, an open-label SPECT/CT (single photon emission computed tomography / computed tomography) study to investigate 99mTc-3PRGD2 SPECT/CT in diagnosis and efficacy evaluation of breast cancer. A single dose of nearly 0.3 mCi/kg body weight 99mTc-3PRGD2 ( ≤ 20 µg 3PRGD2) will be intravenously injected into the patients. Visual and semiquantitative method will be used to assess the whole-body planar and lesions SPECT/CT images. Adverse events will also be observed in the patients.

ELIGIBILITY:
Diagnostic group：

Inclusion Criteria:

* Males and females, ≥20 years old.
* Part of lesion CT and/or 18F-FDG PET/CT and/or MRI and/or Doppler Ultrasound and/or Mammography diagnosis in suspicion of primary or recurrent breast cancer.
* The above cancers will be histologically confirmed or results of histology will be available.

Exclusion Criteria:

* Females planning to bear a child recently or with childbearing potential.
* Known severe allergy.
* Inability to lie still for the entire imaging time because of cough, pain, etc.
* Inability to complete the needed examinations due to severe claustrophobia,radiation phobia, etc.
* Concurrent severe and/or uncontrolled and/or unstable other medical disease that, in the opinion of the Investigator, may significantly interfere with study compliance.

Efficacy evaluation group:

Inclusion Criteria:

* Males and females, ≥20 years old.
* Firstly and definitely diagnose with malignant tumors ,and prepare to chemotherapy (including neoadjuvant chemotherapy) or radiotherapy.
* There are available lesions for assessment during the trial.
* Part of lesion CT and/or 18F-FDG PET/CT and/or MRI and/or Doppler Ultrasound and/or Mammography examination before treatment, the mid tern treatment, post-treatment( three months after the initial treatment) are available.

Exclusion Criteria:

* Females planning to bear a child recently or with childbearing potential.
* Known severe allergy or hypersensitivity to IV radiographic contrast.
* Inability to lie still for the entire imaging time because of cough, pain, etc.
* Inability to complete the needed examinations due to severe claustrophobia, radiation phobia, etc.
* Concurrent severe and/or uncontrolled and/or unstable other medical disease that, in the opinion of the Investigator, may significantly interfere with study compliance.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2016-01; Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Visual Assessment of Breast Lesions in 99mTc-3PRGD2 SPECT/CT Scan | One year
  Visual analysis will be performed by 3 experienced nuclear medicine physicians to observe the the uptake of 99mTc-3PRGD2 on breast lesions. The visual analysis interpreter's degree of suspicion for an abnormality was recorded with use of a 3-point with the following categories: score 1, no abnormal increased uptake; score 2, mildly increased uptake; score 3, definite focal increased uptake. The lesion was considered positive as malignancy if the lesion scored as 2 or higher.
Semiquantitative Assessment of Breast Lesions in 99mTc-3PRGD2 SPECT/CT Scan | One year
  The semiquantitative analysis of the standardized uptake values (SUV) of 99mTc-3PRGD2 SPECT/CT was performed on breast lesion.

SECONDARY OUTCOMES:
Adverse events collection | 5 days
  Adverse events within 5 days after the injection and scanning of the patients will be followed and assessed.
Mammography and/or ultrasound | One year
  Mammography and/or ultrasound will be carried out in breast cancer patients to observe the location and tumor diameter (cm).
18F-FDG PET/CT scan | One year
  18F-FDG PET/CT will be carried out in breast cancer patients to assess the uptake of breast lesions, the axillary lymph node metastasis or distant metastasis and the standardized uptake values (SUVs) of these lesions will be measured.
carbohydrate antigen 153 | One year
  The patients will be required to test level of carbohydrate antigen 153 (CA153, U/L) routinely.

CONTACTS AND LOCATIONS:
Overall Officials: Weibing Miao, MD, Principal Investigator — First Affiliated Hospital of Fujian Medical University
Locations (1):
- Department of Nuclear Medicine, First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Chen Z, Fu F, Li F, Zhu Z, Yang Y, Chen X, Jia B, Zheng S, Huang C, Miao W. Comparison of [99mTc]3PRGD2 Imaging and [18F]FDG PET/CT in Breast Cancer and Expression of Integrin alphavbeta3 in Breast Cancer Vascular Endothelial Cells. Mol Imaging Biol. 2018 Oct;20(5):846-856. doi: 10.1007/s11307-018-1178-y. PMID 29497956